CLINICAL TRIAL: NCT03000361
Title: Motorized Spiral Colonoscopy Trial (MSCT): A First Feasibility Trial
Brief Title: Motorized Spiral Colonoscopy Trial: A First Feasibility Trial
Acronym: MSCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Evangelisches Krankenhaus Düsseldorf (Other)
Collaborators: Olympus (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MSCT
Record Dates: First submitted 2016-12-15; First posted 2016-12-22 (Estimated); Last update posted 2017-08-01 (Actual); Status verified 2017-07

CONDITIONS: Colonoscopy; Safety Issues; Adenoma
Keywords: Colonoscopy; motorized spiral endoscopy; adenoma detection rate
MeSH Terms: conditions — Adenoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Motorized Spiral Colonoscopy (Experimental): Motorized Spiral Colonoscopy (MSC) with the novel motorized spiral endoscope represents a new technology which offers all of the advantageous options of spiral-assisted endoscopy with a faster and less invasive approach
  Interventions: Procedure: Motorized Spiral Colonoscopy

INTERVENTIONS:
Procedure: Motorized Spiral Colonoscopy — For any pathological finding during colonoscopy standard endoscopic techniques, e.g. forceps biopsy, injection, endoscopic mucosal resection, argon plasma coagulation
  Other Names: standard endoscopic interventions (not experimental)

SUMMARY:
The aim of this study is to assess the feasibility and the safety of the Novel Motorized Spiral Endoscope to examine the colon. The study is conceived as proof of concept trial with the primary aim to achieve a cecal intubation rate of at least 90 % according to quality guidelines recommendations. All other clinically relevant quality parameters of standard colonoscopy will be evaluated as secondary aims comparable to our recent trial. This study represents the first clinical evaluation of using a motorized spiral assisted endoscope for examination of the colon with potential advantages for patients in terms of effectiveness and convenience of colonoscopy.

DETAILED DESCRIPTION:
Colonoscopy has been widely accepted for the diagnosis and treatment of colon diseases. Properly performed, colonoscopy is generally safe, accurate, and well-tolerated. Diagnostic colonoscopy is the preferred method to evaluate the colon in most patients with large-bowel symptoms, iron deficiency anemia, abnormal results on radiographic studies of the colon, positive results on colorectal cancer (CRC) screening tests, post-polypectomy and post-cancer resection surveillance, and diagnosis and surveillance in inflammatory bowel disease. In addition, colonoscopy has been introduced for CRC screening in some Western countries e.g. in the United States and Germany. Recent trials showed that screening colonoscopy has a large potential for prevention and early detection of colorectal cancer. Diagnostic colonoscopy is usually combined with endoscopic resection of small and medium sized polyps and flat neoplastic lesions. Patients in whom larger lesions are detected at a diagnostic colonoscopy are usually rescheduled for therapeutic colonoscopy in an appropriate setting.

Quality parameters for colonoscopy were recently reported. In terms of intraprocedural indicators a cecal intubation rate of ≥ 90% for all cases of colonoscopy is widely accepted. Even experienced endoscopists classify up to 10% of colonoscopies as difficult and intubation of the cecum may then be impossible. A recent study evaluated the efficacy and safety of repeating colonoscopy in 520 patients with prior incomplete colonoscopy. Reasons for failure to complete colonoscopy in referring institutions were "looping/redundant colon" in 53.8% of the cases, "sigmoid fixation/angulation" in 38.8%, "both sigmoid angulation and looping colon" in 5.8% of the cases. Issues with sedation caused failures in 1.5% of the patients. Conventional colonoscopy can be difficult in particular in these anatomical variations because pushing the endoscope tends to form loops with limited or no advancement of the tip of the instrument. Techniques like alternating pushing and pulling the endoscope or external compression of the abdomen are used to overcome these limitations. Loop formation and stretching the colon with the adjacent mesenterium as well as external compression are inconvenient or even painful for the patient. In addition these maneuvers prolong the procedural duration. We recently compared the use of ultrathin colonoscopies with standard colonoscope in a randomized trial in terms of cecal intubation rate, level of sedation, amount of propofol needed for sedation, number of external compressions, pain score patient satisfaction and other parameters. The results indicate that these parameters can be well used for evaluation of a new technique of colonoscopy.

Spiral assisted endoscopy is based on a completely different concept of advancing an endoscope by pleating of bowel on the instrumentation shaft by rotation. This technique has been widely used for antegrade enteroscopy. For this purpose a manually rotatable overtube is used through which a thin flexible enteroscope is inserted. The distal end of the overtube contains a raised spiral thread for pleating the small intestine over the overtube. By manually rotating the spiral element the bowel pleats onto the overtube, allowing the operator to access and visualize the more distal portions of the small intestine. Spiral assisted endoscopy has been also approved and evaluated for retrograde enteroscopy via the anal route. It promises advantage for intubation of the cecum and the terminal ileum by its principle of pleating at least parts of the colon with consecutive shortening and less loop formation. These effects should reduce the need for external compression and they may cause less pain for patients. In addition, the spiral should stabilize the position of the colonoscope which is advantageous for careful examination and targeted interventions. Spiral overtube-assisted colonoscopy achieved a success rate of cecal intubation in 92% of 24 patients in whom conventional colonoscopy had failed. However conventional spiral endoscopy is cumbersome to use and requires assistance by a second endoscopist for its appropriate use.

The Novel Motorized Spiral Endoscope represents a new technology which offers all of the advantageous options of spiral-assisted endoscopy with a faster and less invasive approach. The system is similar to other currently marketed endoscopes in that it incorporates a flexible insertion tube, light source, digital imaging, and channels for passing accessories for sample collection or therapeutic interventions. The system is unique in that it incorporates a user-controlled motor contained in the endoscope's handle to rotate a spiral cuff located on the endoscope's insertion tube. Rotation of this cuff, which has soft spiral-shaped "fins", pleats the colon on to the endoscope's insertion tube, thereby allowing rapid and atraumatic access into the colon. The system also includes a display monitor, a motor control unit, device to display measured motor current and signal torque, and a set of foot pedals. It is currently being evaluated in a prospective study in patients with indications for antegrade enteroscopy ("European Novel Motorized Spiral Endoscopy Trial (ENMSET)) in the two centers conducting this study. So far more than 60 patients were successfully examined without major adverse events.

The aim of this study is to assess the feasibility and the safety of the Novel Motorized Spiral Endoscope to examine the colon. The study is conceived as proof of concept trial with the primary aim to achieve a cecal intubation rate of at least 90 % according to quality guidelines recommendations. All other clinically relevant quality parameters of standard colonoscopy will be evaluated as secondary aims comparable to our recent trial. This study represents the first clinical evaluation of using a motorized spiral assisted endoscope for examination of the colon with potential advantages for patients in terms of effectiveness and convenience of colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Screening for colorectal neoplasia
* Surveillance after previous polypectomy/endoscopic mucosal resection (EMR)
* Positive results on colorectal cancer (CRC) screening tests
* Evaluation of clinical symptoms of non overt gastrointestinal bleeding
* Indeterminate iron-deficiency anaemia
* Chronic diarrhoea
* Indeterminate large-bowel symptoms requiring evaluation for colorectal disease

Exclusion Criteria:

* Age under 18 years
* Health status American Society of Anesthesiologists classification (ASA) level ≥ 3
* Pregnancy
* Known coagulopathy (INR≥2.0, Platelets < 70/nl)
* Anti-platelet agents or anticoagulants (other than aspirin) within last 7 days
* History of chronic inflammatory bowel disease
* Previously identified colorectal polyps/lesions with indication for endoscopic resection
* Any medical contraindication to standard colonoscopy
* Any prior abdominal surgery of the mid or lower gastrointestinal tract (except uncomplicated appendectomy)
* Known or suspected bowel obstruction or stenosis
* Known hemorrhoids 3rd degree
* Suspected perforation of the GI tract
* Inability to tolerate sedation for any reason
* Absence of a signed informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-12; Primary Completion 2017-02-01 (Actual); Study Completion 2017-02-01 (Actual)

PRIMARY OUTCOMES:
Cecal intubation rate | 3 days

SECONDARY OUTCOMES:
Ileum intubation rate | 3 days
Procedure time | 3 days
rate of need for external compression | 3 days
  external compression necessary during intervention, yes/no?
adenoma detection rate | 3 days
success rate for removal of polyps | 3 days
amount of propofol needed for sedation | 3 days
maximum level of sedation during procedure | 3 days
  sedation depth assessed by ESGE-guideline, level 1-3
patient satisfaction score | 3 days
  1-10 visual analog scale
adverse event rate | 3 days
maximum pain during procedure | 3 days
  1-10 visual analog scale

CONTACTS AND LOCATIONS:
Overall Officials: Horst Neuhaus, MD, PhD, Principal Investigator — Evangelisches Krankenhaus Duesseldorf, Germany
Locations (1):
- Evangelisches Krankenhaus, Düsseldorf, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Beyna T, Schneider M, Pullmann D, Gerges C, Kandler J, Neuhaus H. Motorized spiral colonoscopy: a first single-center feasibility trial. Endoscopy. 2018 May;50(5):518-523. doi: 10.1055/s-0043-123577. Epub 2017 Dec 18. PMID 29253918